CLINICAL TRIAL: NCT07264621
Title: Adaptive Multi-tiered School-based Prevention to Promote Youth Mental Health and Create Equitable and Sustainable Systems of Care
Brief Title: The University of Oregon ACCESS Project
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001745; 1P50MH139449 (NIH)
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: School Attendance; School Climate; School Engagement; School Exclusion; Externalizing Behavior; Disparities; Teacher-student Relationships; Stress; Emotional Regulation; Depression
Keywords: school-based intervention; family intervention; middle school; SMART trial
MeSH Terms: conditions — Emotional Regulation; Depression

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomization Trial (SMART)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- School-As-Usual (SAU) Only (No Intervention): Students were selected to participate in the study based on meeting attendance and behavioral criteria in 6th grade for Tier 2 or Tier 3 school supports. Students in this arm attended 7th grade at a school in the School-As-Usual condition and therefore did not receive the Tier 1 intervention, ISLA. In addition, in January of 7th grade their school behavior and attendance no longer met criteria for assignment to the Tier 2 intervention, the Family Check-up Online. Thus, students in this arm received neither the ISLA nor FCU-O interventions.
- SAU + FCU Online Only (Experimental): Students were selected to participate in the study based on meeting attendance and behavioral criteria in 6th grade for Tier 2 or Tier 3 school supports. Students in this arm attended 7th grade at a school in the School-As-Usual condition and therefore did not receive the Tier 1 intervention, ISLA. In January of 7th grade their school behavior and attendance continued to meet criteria for assignment to Tier 2 intervention, and thus they received the Family Check-Up Online. In this arm, students' parents were assigned to receive the Family Check-Up Online digital intervention only (without supportive telehealth coaching).
  Interventions: Behavioral: Family Check-Up Online (FCU-O)
- SAU + FCU Online with Telehealth Coaching (Experimental): Students were selected to participate in the study based on meeting attendance and behavioral criteria in 6th grade for Tier 2 or Tier 3 school supports. Students in this arm attended 7th grade at a school in the SAU condition, and therefore did not receive the Tier 1 intervention, ISLA. In January of 7th grade their school behavior and attendance continued to meet criteria for Tier 2 intervention, and thus they received the Family Check-Up Online. In this arm, students' parents were assigned to receive the Family Check-Up Online digital intervention and telehealth coaching to support uptake of FCU content.
  Interventions: Behavioral: FCU-Online with telehealth coaching
- ISLA intervention + FCU Online Only (Experimental): Students were selected to participate in the study based on meeting attendance and behavioral criteria in 6th grade for Tier 2 or Tier 3 school supports. Students in this arm attended 7th grade at a school which implemented the school-wide Tier 1 intervention, ISLA. In January of 7th grade their school behavior and attendance continued to meet criteria for Tier 2 intervention, and thus they received the Family Check-Up Online. In this arm, students' parents were assigned to receive the Family Check-Up Online digital intervention only (without supportive telehealth coaching).
  Interventions: Behavioral: Inclusive Skill-building Learning Approach (ISLA); Behavioral: Family Check-Up Online (FCU-O)
- ISLA intervention+ FCU Online with Telehealth Coaching (Experimental): Students were selected to participate in the study based on meeting attendance and behavioral criteria in 6th grade for Tier 2 or Tier 3 school supports. Students in this arm attended a school which implemented the school-wide Tier 1 intervention, ISLA. In January of 7th grade their school behavior and attendance continued to meet criteria for Tier 2 intervention, and thus they received the Family Check-Up Online. In this arm, students' parents were assigned to receive the Family Check-Up Online digital intervention with telehealth coaching to support uptake of the FCU content.
  Interventions: Behavioral: Inclusive Skill-building Learning Approach (ISLA); Behavioral: FCU-Online with telehealth coaching
- ISLA Intervention Only (Experimental): Students were selected to participate in the study based on meeting attendance and behavioral criteria in 6th grade for Tier 2 or Tier 3 school supports. Students in this arm attended a school which implemented the school-wide Tier 1 intervention, ISLA. In January of 7th grade their attendance and behavior no longer met criteria for Tier 2 intervention. Thus, their parents were not offered the FCU Online digital intervention.
  Interventions: Behavioral: Inclusive Skill-building Learning Approach (ISLA)

INTERVENTIONS:
Behavioral: Inclusive Skill-building Learning Approach (ISLA) — ISLA is a school-wide, multi-component, instructional and restorative alternative to exclusionary discipline that involves universal prevention grounded in positive, preventative classroom strategies for all students, and layers on additional supports for students in need.Derived from the original School-Wide Positive Behavioral Interventions model (SWPBIS) with roots in social learning theory, ISLA emphasizes that behavior is learned through modeling and teaching, and that environmental factors and the quality of teaching practices influence when and how a behavior is likely to occur. The ISLA model emphasizes ongoing training and coaching of classroom-level prevention strategies and practices that teachers use to promote building strong relationships, preventing school disconnectedness, and improving instructional and restorative alternatives to exclusion.
  Arms: ISLA Intervention Only; ISLA intervention + FCU Online Only; ISLA intervention+ FCU Online with Telehealth Coaching
Behavioral: Family Check-Up Online (FCU-O) — The Family Check-Up Online is a digital intervention that includes an assessment, computer-generated feedback, and intervention modules that focus on improving family relationships and parenting skills in order to reduce child mental health problems and to improve child self-regulation. These modules include Healthy Behaviors for Stressful Times, Positive Parenting, Rules and Consequences, Supporting School Success, and Communication.
  Arms: ISLA intervention + FCU Online Only; SAU + FCU Online Only
Behavioral: FCU-Online with telehealth coaching — This intervention is the Family Check-Up Online plus telehealth support from a parenting coach. The Family Check-Up Online is a digital intervention that includes an assessment, computer-generated feedback, and intervention modules that focus on improving family relationships and parenting skills in order to reduce child mental health problems and to improve child self-regulation. These modules include Healthy Behaviors for Stressful Times, Positive Parenting, Rules and Consequences, Supporting School Success, and Communication. A coach based at the child's school meets with caregivers via telehealth modality to provide motivation and to help caregivers tailor the content of the modules to their specific child and family's needs.
  Arms: ISLA intervention+ FCU Online with Telehealth Coaching; SAU + FCU Online with Telehealth Coaching

SUMMARY:
The goal of this clinical trial is to learn if two behavioral interventions work to reduce office disciplinary referrals, improve attendance, and reduce depression and anxiety in 7th grade students. This project combines two evidence-based programs-the Inclusive Skill-building Learning Approach (ISLA) for school-wide discipline reform and the Family Check-Up Online (FCU-O) for family-centered support-in an adaptive design to examine the unique and additive effects of these interventions on these child behavior outcomes.

The main questions it will answer are:

1. What is the relative efficacy of ISLA vs. School-as-Usual?
2. What is the optimal sequencing of these interventions?
3. Which overall sequence of intervention strategies was most effective?

Researchers will compare 6 combinations of these interventions to see which combination and sequencing provides the best student outcomes.

School personnel participating in the project will be trained to implement the two interventions at their school. They will answer surveys in the fall, winter, and spring of their year of participation. Parent and Youth participants will complete surveys at baseline and then again 6 months and 12 months later.

DETAILED DESCRIPTION:
In the past decade, youth mental health and behavior concerns have been some of the most significant challenges in schools, exacerbated by the COVID-19 pandemic. A high percentage of adolescents experience mental health distress, but only a fraction of them recieve adequate services, especially in underserved communities. School-based services face barriers such as limited funding, staffing shortages, and a lack of evidence-based programming. Mental health issues are driven by a combination of individual and systemic risk factors, including inequitable school policies, caregiver stress, and family history of mental health disorders. Youth from minoritized backgrounds face higher stressors, further impacting their mental health. Due to the complexity and depth of these issues, an approach that intervenes on a school- and family-level could show significant reduction in mental health and behavioral concerns which would otherwise precipitate into a lifetime of cascading negative outcomes.

Effective strategies that can aid in this youth mental health epidemic include family-centered treatments and school-wide programs to reduce exclusionary discipline practices, which disproportionately affect marginalized students and contribute to the school-to-prison pipeline. Family engagement in mental health interventions has shown positive, long-term effects, but participation rates remain low, with most school programs focusing on individual students rather than families.

This project aims to highlight the importance of embedding mental health services in schools by way of providing schools with equitable skill-building supports to improve student social and behavioral problem-solving, as well as providing families with a brief, strengths-based, digital health intervention for families to reduce mental health and behavioral concerns by improving emotional regulation and family relationships. Digital health interventions, like web-based programs, offer a promising solution to reach underserved families and students. This project combines two evidence-based programs-the Inclusive Skill-building Learning Approach (ISLA) for school-wide discipline reform and the Family Check-Up Online (FCU-O) for family-centered support-in an adaptive design. Integrating a family-centered intervention that promotes positive and nurturing familial relationships with a systemic intervention that addresses inequitable discipline practices in schools provides a promising and innovative approach for reducing the youth mental health crisis across multiple systems, including home, school, and communities. This approach aims to reduce mental health issues by addressing both school and family dynamics. The project evaluates the effectiveness and sustainability of these interventions using a multi-level model and randomized trials.

ELIGIBILITY:
School Inclusion Criteria:

* The middle school must be located in Oregon and serve a population with high levels of NIH-defined health disparity; and
* The middle school must have a history of collaboration with the National PBIS Technical Assistance Center or the Northwest PBIS network.

School Staff Inclusion Criteria:

* School staff must be employed by a participating middle school; and
* School staff must be willing and interested in receiving training and support throughout implementation

Family Inclusion Criteria:

* The target child must attend a middle school which has been randomly assigned to receive the ISLA intervention or School-as-Usual;
* The target child must be in 7th grade and between the ages of 11 and 14;
* The caregiver must be the parent or legal guardian of the target child;
* The target child must exhibit at least one of the following risk factors during the prior academic year (6th grade):
* 2 or more office discipline referrals;
* poor attendance, i.e., missing 2 more school days per month; and
* The caregiver must have a smartphone with text messaging capability, access to email and internet.

Family Exclusion Criteria:

Families will be excluded from the study if:

* the caregiver is unable to read in either English or Spanish;
* either member of the parent-child dyad chooses not to participate (i.e., both members of the dyad need to consent/ assent); or
* the family is already participating in another study at the University of Oregon's Prevention Science Institute.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Child Depression (Parent Report) | baseline, 6 months, 12 months
  Parents report on their child's depression using the eight item PHQ-8. Parents are asked to indicate how often their child has experienced symptoms over the last two weeks using a 4-pt Likert scale: 0 =not at all, 1=several days, 2=more than half the days, 3= nearly every day. Scores for individual items are summed together. Higher scores indicate greater child depression.
Change from Baseline in Child Depression (Student Report) | baseline, 6 months, 12 months
  Students report on their symptoms of depression using the eight item PHQ-8. Students are asked to indicate how often they have experienced symptoms over the last two weeks using a 4-pt Likert scale: 0 =not at all, 1=several days, 2=more than half the days, 3= nearly every day. Scores for individual items are summed together. Higher scores indicate greater child depression.
Change from Baseline in Child Anxiety (Parent Report) | baseline, 6 months, 12 months
  Parents report on their child's anxiety using the 7 item GAD-7. Parents are asked to indicate how often their child has experienced symptoms over the past 2 weeks using a 4-pt Likert scale: 0= not at all, 1=several days, 2=more than half the days, and 3= nearly every day. Ratings of the 7 items are summed together. Higher scores indicate greater child anxiety.
Change from Baseline in Child Anxiety (Student Report) | baseline, 6 months, 12 months
  Students report on their symptoms of anxiety using the 7 item GAD-7. Students are asked to indicate how often they have experienced symptoms over the past 2 weeks using a 4-pt Likert scale: 0= not at all, 1=several days, 2=more than half the days, and 3= nearly every day. Ratings of the 7 items are summed together. Higher scores indicate greater child anxiety.
Change from Baseline in Student Problem Behaviors (Parent Report) | baseline, 6 months, 12 months
  The Strengths and Difficulties Questionnaire (SDQ; Goodman 1997) is a 25-item behavioral screening questionnaire about psychosocial problems for youth, and includes competencies or strengths in addition to assessing problems. The SDQ is equally divided across five scales measuring emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior. Parents are provided statements and asked to indicate how true each statement has been for their child over the past 6 months using a 3-pt Likert scale: 0=Not True, 1=Somewhat True, and 2=Certainly True. Ratings are summed, and higher scores indicate more problem behavior.
Change from Baseline in Student Problem Behaviors (Student Report) | baseline, 6 months, 12 months
  The Strengths and Difficulties Questionnaire (SDQ; Goodman 1997) is a 25-item behavioral screening questionnaire about psychosocial problems for youth, and includes competencies or strengths in addition to assessing problems. The SDQ is equally divided across five scales measuring emotional symptoms, conduct problems, hyperactivity-inattention, peer problems, and prosocial behavior. Students are provided statements and asked to indicate how true each statement has been for them over the past 6 months using a 3-pt Likert scale: 0=Not True, 1=Somewhat True, and 2=Certainly True. Ratings are summed, and higher scores indicate more problem behavior.
Change from Baseline in School Climate (Student Report) | baseline, 6 months, 12 months
  The School Climate Survey: Secondary (SCS-S) is a 36-item school climate rating scale (Center on PBIS, 2022) intended to obtain middle and high school student perception ratings of school climate. It has 8 subscales: school connectedness, peer social support, adult social support, cultural acceptance, social/ civic learning, physical environment, school safety, and order and discipline. Respondents use a 4-point Likert scale: 1=Strongly Disagree, 2 = Somewhat Disagree, 3 = Somewhat Agree, and 4 = Strongly Agree. To compute the overall school climate score, item responses are summed and then divided by the total number of items. Higher overall scores reflect a more positive sense of the school environment.
Change from Baseline in School Climate (Teacher Report) | Fall, Winter, and Spring of one academic year (e.g., baseline, 6 months, 10 months)
  The School Climate Survey: School Personnel (Center on PBIS, 2022) includes 29 items and 5 subscales, including staff connectedness, structure for learning, school safety, physical environment, peer and adult relations, and parent involvement. School personnel rate items with a four-point Likert scale: 1=Strongly Disagree, 2=Somewhat Disagree, 3=Somewhat Agree, and 4=Strongly Agree. To compute the overall school climate score, item responses are summed and then divided by the total number of items. Higher overall scores reflect a more positive sense of the school environment.
Change from Baseline in Number of ODRs, In-School Suspensions, and Out-of-School Suspensions (School-Level) | Fall, winter, and spring of two academic years (baseline, 6 months, 9 months, 12 months, 18 months, 21 months)
  The number of office disciplinary referrals (ODRs), in-school (ISS), and out-of-school suspensions (OSS) will be gleaned from school records and aggregated at the school-level.
Change from Baseline in Number of ODRs, In-School Suspensions, and Out-of-School Suspensions (Student-Level) | baseline, 12 months
  The number of office disciplinary referrals (ODRs), in-school (ISS), and out-of-school suspensions (OSS) received by participating students will be gleaned from school records and recorded at the student-level for two academic years (6th grade and 7th grade).
Change from Baseline in Number of Days Absent from School (Student-Level) | Time Frame: baseline, 12 months
  The number of days that participating students were absent from school will be gleaned from school records and recorded at the student-level for two academic years (6th grade and 7th grade).

CONTACTS AND LOCATIONS:
Overall Officials: Beth Stormshak, PhD, Principal Investigator — University of Oregon; Rhonda Nese, PhD, Principal Investigator — University of Oregon
Locations (13):
- United States (13):
  - Lincoln Middle School, Cottage Grove, Oregon
  - Monroe Middle School, Eugene, Oregon
  - Kelly Middle School, Eugene, Oregon
  - Madison Middle School, Eugene, Oregon
  - Arts & Technology Academy, Eugene, Oregon
  - Kennedy Middle School, Eugene, Oregon
  - Roosevelt Middle School, Eugene, Oregon
  - Spencer Butte Middle School, Eugene, Oregon
  - Cal Young Middle School, Eugene, Oregon
  - Briggs Middle School, Springfield, Oregon
  - Hamlin Middle School, Springfield, Oregon
  - Agnes Stewart Middle School, Springfield, Oregon
  - Thurston Middle School, Springfield, Oregon

IPD SHARING:
Plan to Share IPD: Yes
De-identified, final research data generated in the research activities, along with metadata, descriptors, and protocols, will be shared with the broader scientific community. Material to be shared include detailed protocols and recommendations for schools to increase the health and wellbeing of middle schoolers. Researchers outside of the ACCESS Center will have access to a standard de-identified, individual-level dataset held to the same standard as that established by the HIPAA Privacy Rule. General documentation will be available without cost in the form of PDF files. Potentially identifying fields as defined in the HIPAA Privacy Rule will not be released to outside researchers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After completion of the project funding period, de-identified, final research data generated in the research activities, along with metadata, descriptors, and protocols, will be shared with the broader scientific community through dissemination efforts and uploads to the NIMH Data Archive.
Access Criteria: External researcher requests for de-identified individual-level data must be accompanied by a signed Data Use Agreement, and researchers must document that they are working under an institution with a Federal Wide Assurance (FWA).To optimize usage of the data, the website at the University of Oregon's ACCESS Center will provide clear instructions for accessing the data.
URL: https://blogs.uoregon.edu/psiaccesscenter/